CLINICAL TRIAL: NCT06331455
Title: Treatment of Pulmonary SUlcus, Pancoast and Chest Wall Non-small Cell Lung Cancer
Brief Title: Treatment of Pulmonary SUlcus, Pancoast and Chest Wall Non-small Cell Lung Cancer Employing Radiation, Immuno-oncology and Resection
Acronym: SUPER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marc de Perrot (Other)
Collaborators: Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor-Investigator, Marc de Perrot, Thoracic Surgeon, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-5501
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer Patients; Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: This is a multi-centre, phase 2 trial in patients with T2b-3N0-1M0 NSCLC evaluating the biologic efficacy of NORT-Durvalumab administered prior to surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant NORT-Durvalumab (Experimental): administration of non-ablative oligofractionated radiation therapy using 12 Gy in 3 fractions in combination with two doses of durvalumab (1500 mg IV) prior to surgery.
  Interventions: Drug: Durvalumab; Radiation: Non-ablative oligofractionated radiation (NORT)

INTERVENTIONS:
Drug: Durvalumab — Two doses of durvalumab (1500 mg IV)
Radiation: Non-ablative oligofractionated radiation (NORT) — 12 Gy of Radiation in 3 fractions

SUMMARY:
The SUPER trial is a prospective Phase II trial. It is designed for patients with stage 2 or 3 non-small cell lung cancer (NSCLC) prior to surgery.

Patients who are enrolled in this trial will receive combination of Non-ablative oligofractionated radiation (NORT) and two cycles of Durvalumab, an immunotherapy drug before their surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Age > 18 years at time of study entry.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Body weight >30 kg
5. Adequate normal organ and marrow function as defined below Hemoglobin ≥9.0 g/dL Absolute neutrophil count (ANC) ≥1.0 × 10^9/L Platelet count ≥75 × 10^9/L Serum bilirubin in normal range with the exception of Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal

   Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min)=Weight (kg) x (140 - Age) / 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min)=Weight (kg) x (140 - Age) x 0.85 / 72 x serum creatinine (mg/dL)
6. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
7. Must have a life expectancy of at least 12 weeks
8. Tumor amenable to biopsy
9. Patients with NSCLC stage IIB to IIIB.
10. PD-L1 positive tumors defined by tumor proportion score (TPS) >1%
11. Patient suitable for surgery and combined modality therapy in the opinion of the investigator.
12. Complete R0 resection of the primary tumor and involved lymph nodes is anticipated based on the clinical staging and radiological evaluation according to the baseline pre-treatment imaging.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 8 weeks before enrollment
2. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
3. Known oncogenic driver mutations such as EGFR mutant or ALK mutant
4. The presence of N3 disease in the contralateral mediastinum, contralateral hilum, or contralateral supraclavicular lymph node confirmed histologically.
5. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Sponsor.

   Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the StudySponsor.
6. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
7. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
8. History of allogenic organ transplantation.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   Patients with vitiligo or alopecia Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement Any chronic skin condition that does not require systemic therapy Patients without active disease in the last 5 years may be included but only after consultation with the Study Sponsor Patients with celiac disease controlled by diet alone
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
11. History of another primary malignancy except for:

    Malignancy treated with curative intent that does not require treatment, nor anticipated to require treatment for the duration of the study, and in the opinion of the investigator would not pose a risk of increased toxicity, or difficulty to follow the protocol and assess study endpoints Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease Adequately treated carcinoma in situ without evidence of disease
12. History of leptomeningeal carcinomatosis, malignant pleural effusion or distant metastasis (M1)
13. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry
14. History of active primary immunodeficiency
15. Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
16. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
18. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
19. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
20. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
21. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
22. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4:

    Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.

    All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.

    Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE:

    Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.

    Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
23. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To Measure CD8 TILs density & Major Pathological Response (MPR) | 5-6 weeks post treatment
  1. The proportion of patients achieving MPR after neoadjuvant therapy
  2. The proportion of patients doubling the CD8 TILs density after neoadjuvant therapy.

SECONDARY OUTCOMES:
To explore the efficacy and safety of NORT-durvalumab | 12 weeks post surgery
  1. The proportion of patients achieving pCR after neoadjuvant therapy
  2. The proportion of patients with grade 3, 4 or 5 toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Marc de Perrot, MD, FRCSC, Principal Investigator — UHN - Toronto General Hopsital
Locations (1):
- Toronto General Hospital, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No